CLINICAL TRIAL: NCT00317642
Title: A Phase III Randomized, Double-blind, Controlled Study Comparing Clofarabine and Cytarabine Versus Cytarabine Alone in Adult Patients 55 Years and Older With Acute Myelogenous Leukemia (AML) Who Have Relapsed or Are Refractory After Receiving up to Two Prior Induction Regimens
Brief Title: A Study of Clofarabine and Cytarabine for Older Patients With Relapsed or Refractory Acute Myelogenous Leukemia (AML)(CLASSIC I)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLO34100405; 2008-001043-19 (EudraCT Number)
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Results first posted 2011-09-15 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Acute Myelogenous Leukemia
Keywords: acute myelogenous leukemia; acute myeloid leukemia; relapsed AML; refractory AML; clofarabine; cytarabine; CLO341; clolar
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine; Dosage Forms; Cytarabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clofarabine (IV formulation) and cytarabine (Experimental): Participants received clofarabine (40 mg/m^2) administered as a 1-hour infusion followed 3 hours later (from end of infusion) by cytarabine 1 g/m^2 administered as a 2-hour infusion. Participants could receive up to 3 cycles of treatment (induction, re-induction, and consolidation)
  Complete induction cycle = 5 consecutive days of treatment
  Re-induction cycle = 5 consecutive days of treatment at the original or modified dose
  Consolidation cycle = 4 consecutive days of treatment at the original or modified dose
  Interventions: Drug: clofarabine (IV formulation); Drug: cytarabine
- placebo and cytarabine (Experimental): Participants received placebo administered as a 1-hour infusion followed 3 hours later (from end of infusion) by cytarabine 1 g/m^2 administered as a 2-hour infusion. Patients could receive up to 3 cycles of treatment (induction, re-induction, and consolidation)
  Interventions: Drug: placebo; Drug: cytarabine

INTERVENTIONS:
Drug: clofarabine (IV formulation) — clofarabine (IV formulation) infusion 40mg/m^2 / day up to 3 cycles
  Other Names: Clolar®; Evoltra®
  Arms: clofarabine (IV formulation) and cytarabine
Drug: placebo — placebo (sodium Chloride) 1-hour IV infusion
  Arms: placebo and cytarabine
Drug: cytarabine — cytarabine IV infusion 1g/m^2/day for up to 3 cycles

SUMMARY:
Clofarabine (injection) is approved by the Food and Drug Administration (FDA) for the treatment of pediatric patients 1 to 21 years old with relapsed acute or refractory lymphoblastic leukemia (ALL) who have had at least 2 prior treatment regimens.

There is no recommended standard treatment for relapsed or refractory acute myelogenous leukemia in older patients. Cytarabine is the most commonly used drug to treat these patients. This study will determine if there is benefit by combining clofarabine with cytarabine. Patients will be randomized to receive up to 3 cycles of treatment with either placebo in combination with cytarabine or clofarabine in combination with cytarabine. Randomization was stratified by remission status following the first induction regimen (no remission [i.e., CR1 = refractory] or remission <6 months vs CR1 = remission ≥6 months). CR1 is defined as remission after first pre-study induction regimen. The safety and tolerability of clofarabine in combination with cytarabine and cytarabine alone will be monitored throughout the study.

DETAILED DESCRIPTION:
After screening and eligibility assessment, patients were randomized (in a 1:1 ratio) to receive either clofarabine or matching placebo, in addition to cytarabine. Randomization was stratified by remission status following the first induction regimen (CR1): no remission [i.e., CR1 = refractory] or remission <6 months vs remission ≥6 months. During randomization by interactive voice response system (IVRS), there were 10 participants misclassified to the CR1 <6 months stratum and 12 participants misclassified to CR1 ≥6 months stratum. The error did not affect the participants' treatment, only the stratification. Due to the misclassification, outcomes that used strata in their analysis were analyzed twice: once with the 'randomized stratification' which includes the misclassification and once with the 'calculated stratification' in which participants appear in the 'correct' strata.

Two clinical study reports were written for this study.

1. Clinical study report dated 7 April 2011 includes the entire treatment period of all participants plus much of the follow-up. At that time, 33 participants in the Clofarabine+cytarabine group and 29 participants in the placebo+cytarabine group were still being follow-up post treatment. Results were reported on clinicaltrials.gov in August 2011. Outcomes that used strata reported the 'calculated strata' on clinicaltrials.gov.
2. Clinical study report dated 9 July 2012 includes all patient treatment experience plus all long-term follow-up (a minimum of 2 years from the end of treatment or until the patient died). The study was completed at that time. Outcomes that used strata reported the 'randomized strata' on clinicaltrials.gov. AE records on clinicaltrials.gov reflect the final database.

Outcomes that changed between the two clinical study reports due to the additional long-term follow-up data are reported twice on clinicaltrials.gov (once from each clinical study report) and the appropriate report date is included in the outcome description. Outcomes from the 9 July 2012 report represent more complete data.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Acute Myelogenous Leukemia (AML) according to World Health Organization (WHO) classification
* Relapsed after receiving up to 2 prior induction regimens (i.e. first or second relapse)or are refractory to not more than one prior combination chemotherapy induction regimen
* Be ≥ 55 years of age
* Have an Eastern Cooperative Oncology Group (ECOG) score of 0-2
* Be able to comply with study procedures and follow-up examinations
* Be nonfertile or agree to use birth control during the study through the end of treatment visit and for at least 90 days after the last dose of study drug
* Have adequate liver and renal function as indicated by certain laboratory values

Exclusion Criteria:

* Received previous treatment with clofarabine
* Received bolus, intermediate or high-dose cytarabine as induction therapy unless certain remission criteria are met
* Have received a hematopoietic stem cell transplant (HSCT) within the previous 3 months
* Have moderate or severe graft versus host disease (GVHD), whether acute or chronic
* Are receiving any other chemotherapy or investigational therapy. Patients must have been off prior AML therapy for at least 2-6 weeks prior to entering study.
* Have a psychiatric disorder that would interfere with consent, study participation, or follow-up
* Have an active, uncontrolled infection
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system
* Have been diagnosed with another malignancy, unless disease-free for at least 5 years; patients with treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed; patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease are eligible if hormonal therapy has been initiated or the malignancy has been surgically removed.
* Have clinical evidence suggestive of central nervous system (CNS) involvement with leukemia unless lumbar puncture confirms absence of leukemic blasts in the cerebrospinal fluid(CSF)
* Known HIV positivity
* Are pregnant or lactating

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2006-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (57):
- United States (41):
  - Mayo Clinical Hospital, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Arkansas Cancer Research Center, Little Rock, Arkansas
  - Scripps Cancer Center, La Jolla, California
  - UCLA School of Medicine, Los Angeles, California
  - University of Southern California, Kenneth Norris Cancer Center, Los Angeles, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - University of Colorado Health Science Center, Aurora, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - Louisiana State University Health Science Center, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Josephine Ford Cancer Center, Detroit, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Center, Buffalo, New York
  - Mt. Sinai School of Medicine, New York, New York
  - New York Medical Center, Valhalla, New York
  - Mecklenburg Medical Group, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Simmons Comprehensive Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - West Virginia University Hospitals, Mary Babb Randolph Cancer Center, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Juravinski Cancer Center, Hamilton, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
- France (6):
  - Service Maladies du Sang, CHU Angers, Angers
  - Hopital Claude Huriez CHRU de Lille, Lille
  - Hopital Edouard Herriot, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Hotel Dieu, Nantes
  - Hopital Purpan, Toulouse
- Germany (3):
  - Medizinische Hochschule Hannover, Zentrum fur Innere Medizin, Abt. Haematologie / Onkologie, Hanover
  - Medizinische Klinik der Technischen, Universität München, Munich
  - Universitatsklinikum Ulm, Ulm
- Italy (4):
  - Ospedali Riuniti Bergamo, Bergamo
  - A.O Ospedale Niguarda Ca'Granda, Milan
  - N.O. San Gerardo, Monza
  - Azienda Ospedaliera "Antonio Cardarelli", Napoli

REFERENCES:
- [Result] Clofarabine + Ara-c improves response rates and event-free survival, not overall survival, in older patients with relapsed/refractory AML compared to Ara-c alone: Updated CLASSIC I study results. H.M. Kantarjian, M. Wetzler, D. Rizzieri, G. J. Schiller, M. H. Jagasia, R. K. Stuart, S. Ganguly, D. Avigan, M. Craig, R. Collins, M. B. Maris, T. Kovacsovics, S. Goldberg, K. Seiter, P. Hari, J. Greiner, N. Vey, C. Recher, F. Ravandi, E.S. Wang, S. Eckert, D. Huebner and S. Faderl. Haematologica - 16th Congress of EHA Abstracts. 2011; 96(S2): 196.
- [Result] Clofarabine plus cytarabine compared to cytarabine alone in older patients with relapsed or refractory (R/R) acute myelogenous leukemia (AML): Results from the phase III CLASSIC 1 trial. S. Faderl, M. Wetzler, D. Rizzieri, G. J. Schiller, M. H. Jagasia, R. K. Stuart, S. Ganguly, D. Avigan, M. Craig, R. Collins, M. B. Maris, T. Kovacsovics, S. Goldberg, K. Seiter, P. Hari, F. Ravandi, E. S. Wang, S. Eckert, D. Huebner, and H. Kantarjian JCO - ASCO Meeting Abstracts. 2011; 29:6503.
- [Result] Faderl S, Wetzler M, Rizzieri D, Schiller G, Jagasia M, Stuart R, Ganguly S, Avigan D, Craig M, Collins R, Maris M, Kovacsovics T, Goldberg S, Seiter K, Hari P, Greiner J, Vey N, Recher C, Ravandi F, Wang ES, Vasconcelles M, Huebner D, Kantarjian HM. Clofarabine plus cytarabine compared with cytarabine alone in older patients with relapsed or refractory acute myelogenous leukemia: results from the CLASSIC I Trial. J Clin Oncol. 2012 Jul 10;30(20):2492-9. doi: 10.1200/JCO.2011.37.9743. Epub 2012 May 14. PMID 22585697
- [Result] Ganguly S, Kantarjian HM, Wetzler M, Rizzieri D, Schiller G, Jagasia M, et al. Subsequent hematopoietic stem cell transplantation (HSCT) associated with longer survival in patients with relapsed/refractory (R/R) acute myelogenous leukemia (AML) after Clo+Ara-C or Ara-C alone: a landmark analysis from the CLASSIC I trial. Biol Blood Marrow Transplant 2012;18(2Suppl):S211-S212.
- [Result] Ganguly S, Kantarjian HM, Wetzler M, Rizzieri D, Schiller G, Jagasia M, et al. Subsequent HSCT in the CLASSIC I Study Associated with Longer Survival in Patients With Relapsed/Refractory AML After Clo+Ara-C Or Ara-C Alone: A Landmark Analysis. Haematologica - 17th Congress of EHA Abstracts. 2012; 97(s1):32

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 352 patients screened and 326 randomized, 163 to each treatment group. One participant withdrew after being randomized to the Placebo and Cytarabine Group and was excluded from efficacy analysis.
Groups:
- Clofarabine (IV Formulation) and Cytarabine: Participants received clofarabine 40 mg/m^2 administered as a 1-hour intravenous (IV) infusion, followed 3 hours later (from end of infusion) by cytarabine 1 g/m^2 administered as a 2-hour IV infusion for 5 days (induction and re-induction) or 4 days (consolidation). Participants could receive up to 3 cycles of treatment: induction, re-induction (if the participant had not achieved remission following induction but hematological improvement was noted), and consolidation.
- Placebo and Cytarabine: Participants received placebo (sodium chloride) administered as a 1-hour IV infusion, followed 3 hours later (from end of infusion) by cytarabine 1 g/m^2 administered as a 2-hour IV infusion for 5 days (induction and re-induction) or 4 days (consolidation). Participants could receive up to 3 cycles of treatment: induction, re-induction, and consolidation.
Period: Overall Study
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine
Started | 163 | 163
Full Analysis Set | 162 (AML Centrally Confirmed) | 158 (AML Centrally Confirmed)
Received >= 1 Study Drug (Safety Set) | 161 | 155
Completed | 41 (achieved remission and completed consolidation) | 28 (achieved remission and completed consolidation)
Not Completed | 122 | 135
Not completed — Not Received Either Study Drug | 1 | 3
Not completed — Physician Decision | 15 | 7
Not completed — Participant declined treatment | 14 | 3
Not completed — Adverse Event | 17 | 5
Not completed — Treatment Failure | 56 | 102
Not completed — Disease Recurrence | 1 | 2
Not completed — Death | 14 | 7
Not completed — Not Continue to Consolidation | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Referred For Transplantation | 1 | 0
Not completed — AML Not Centrally Confirmed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine | Total
Number analyzed (Participants) | 162 | 158 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (6.36) | 67.1 (5.82) | 67.0 (6.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 57 | 105
  Male | 114 | 101 | 215
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 153 | 152 | 305
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 11 | 18
  White | 150 | 142 | 292
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Height (cm) [Mean (Standard Deviation); unit: centimeter] | 171.5 (10.27) | 170.5 (8.92) | 171.0 (9.62)
Weight(kg) [Mean (Standard Deviation); unit: kg] | 81.21 (17.862) | 83.03 (17.281) | 82.11 (17.574)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.941 (0.2383) | 1.959 (0.2338) | 1.950 (0.2359)
Eastern Cooperative Oncology Group Performance Status [Number; unit: Participants] — Eastern Cooperative Oncology Group Performance Status (ECOG PS) is a scale ranging from 0-5, with 0 (fully active); 1 (capable of light work); 2 (no work but all self-care); 3 (limited self-care); 4 (completely disabled); 5 (dead).
  Participants
    ECOG 0 | 57 | 48 | 105
    ECOG 1 | 79 | 92 | 171
    ECOG 2 | 26 | 18 | 44
Karyotype [Number; unit: participants] — Favorable karyotype was defined as any abnormality of chromosome 16; Intermediate karyotype was defined as normal (no abnormalities); Unfavorable karyotype was defined as any other abnormality
  participants
    Favorable | 1 | 0 | 1
    Intermediate | 65 | 84 | 149
    Unfavorable | 86 | 70 | 156
    Not Assessed | 8 | 3 | 11
    unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival - Overall and by Calculated Strata (CSR 7-April-11)
Description: Overall survival (OS) for the Full Analysis Set (FAS) and for the 2 calculated strata. OS was defined as the number of months from date of randomization until date of death due to any cause.
Time Frame: Day 1 (randomization) up to approximately 4 years
Population: Full Analysis Set (FAS)-all randomized participants whose baseline AML diagnosis was centrally confirmed. Strata are calculated according to duration of the first remission based on case report forms (CRF) data and do not include the IVRS mistakes. One participant's strata (placebo group) could not be calculated so the participant was excluded.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Clofarabine (IV Formulation) and Cytarabine (FAS); Clofarabine and Cytarabine - In Stratum < 6 Months; Clofarabine and Cytarabine In Stratum >= 6 Months: Participants received clofarabine 40 mg/m^2 administered as a 1-hour intravenous (IV) infusion, followed 3 hours later (from end of infusion) by cytarabine 1 g/m^2 administered as a 2-hour IV infusion for 5 days (induction and re-induction) or 4 days (consolidation). Participants could receive up to 3 cycles of treatment: induction, re-induction (if the participant had not achieved remission following induction but hematological improvement was noted), and consolidation.
- Placebo and Cytarabine (FAS); Placebo and Cytarabine - In Stratum < 6 Months; Placebo and Cytarabine In Stratum >= 6 Months: Participants received placebo (sodium chloride) administered as a 1-hour IV infusion, followed 3 hours later (from end of infusion) by cytarabine 1 g/m^2 administered as a 2-hour IV infusion for 5 days (induction and re-induction) or 4 days (consolidation). Participants could receive up to 3 cycles of treatment: induction, re-induction, and consolidation.
Arm/Group | Clofarabine (IV Formulation) and Cytarabine (FAS) | Placebo and Cytarabine (FAS) | Clofarabine and Cytarabine - In Stratum < 6 Months | Placebo and Cytarabine - In Stratum < 6 Months | Clofarabine and Cytarabine In Stratum >= 6 Months | Placebo and Cytarabine In Stratum >= 6 Months
Number analyzed (Participants) | 162 | 157 | 88 | 83 | 74 | 74
months | 6.6 [5.1 to 9.3] | 6.4 [4.7 to 7.3] | 5.1 [3.5 to 8.7] | 5.5 [4.1 to 7.2] | 8.7 [5.3 to 11.1] | 7.2 [4.6 to 8.9]
Statistical Analysis 1: Comparison: Clofarabine (IV Formulation) and Cytarabine (FAS) vs Placebo and Cytarabine (FAS); Full Analysis Set (FAS) population; Test type: Superiority or Other; p = 0.9951, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.78 to 1.28]
Statistical Analysis 2: Comparison: Clofarabine and Cytarabine - In Stratum < 6 Months vs Placebo and Cytarabine - In Stratum < 6 Months; Participants stratified by calculated strata remission after first pre-study induction regimen (CR1) < 6 months; Test type: Superiority or Other; p = 0.4674, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.81 to 1.57]
Statistical Analysis 3: Comparison: Clofarabine and Cytarabine In Stratum >= 6 Months vs Placebo and Cytarabine In Stratum >= 6 Months; Participants stratified by calculated strata CR1>= 6 months; Test type: Superiority or Other; p = 0.3963, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.58 to 1.24]

2. Secondary Outcome: Best Response Per Independent Response Review Panel (IRRP) Assessment - Overall and by Calculated Strata (CSR 7-April-11)
Description: Percentage of participants whose best response was assessed by the IRRP as complete remission (CR) or complete remission with incomplete peripheral blood count recovery (CRi) using the revised International Working Group for Response Criteria (Cheson 2003).
  CR is defined on morphologic criteria at a single response assessment:
  * a bone marrow aspirate or biopsy of <5% blasts, with evidence of normal hematopoiesis;
  * absence of Auer rods in the blasts that are present;
  * absence of extramedullary disease;
  * absence of a unique phenotype determined at the pretreatment specimen, as assessed by immunophenotyping;
  * only rare evidence of circulating blasts. If present, evidence of a regenerating bone marrow;
  * recovery of peripheral counts (platelets ≥100*10^9/L and absolute neutrophil count (ANC) ≥1.0*10^9/L).
  CRi met all criteria for CR except for either residual neutropenia (ANC <1.0*10^9/L) or thrombocytopenia (platelet count <100*10^9/L).
Time Frame: Day 12 up to approximately 6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine | Clofarabine and Cytarabine - In Stratum < 6 Months | Placebo and Cytarabine - In Stratum < 6 Months | Clofarabine and Cytarabine In Stratum >= 6 Months | Placebo and Cytarabine In Stratum >= 6 Months
Number analyzed (Participants) | 162 | 157 | 88 | 83 | 74 | 74
percentage of participants
  Overall Remission (CR + CRi) | 46.9 | 22.9 | 45.5 | 22.9 | 48.6 | 23.0
  Complete Remission (CR) | 35.2 | 17.8 | 33.0 | 18.1 | 37.8 | 17.6
  CR with incomplete blood count recovery (CRi) | 11.7 | 5.1 | 12.5 | 4.8 | 10.8 | 5.4
Statistical Analysis 1: Comparison: Clofarabine (IV Formulation) and Cytarabine vs Placebo and Cytarabine; Full Analysis Set (FAS) population - overall remission (OR); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Clofarabine (IV Formulation) and Cytarabine vs Placebo and Cytarabine; Full Analysis Set (FAS) population - Complete Remission (CR); Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Clofarabine and Cytarabine - In Stratum < 6 Months vs Placebo and Cytarabine - In Stratum < 6 Months; Participants stratified by calculated strata - CR1 <6 months [Overall Remission (CR+CRi)]; Test type: Superiority or Other; p = 0.0022, Fisher Exact
Statistical Analysis 4: Comparison: Clofarabine and Cytarabine In Stratum >= 6 Months vs Placebo and Cytarabine In Stratum >= 6 Months; Participants stratified by calculated strata - CR1 >=6 months [Overall Remission (CR+CRi)]; Test type: Superiority or Other; p = 0.0019, Fisher Exact
Statistical Analysis 5: Comparison: Clofarabine and Cytarabine - In Stratum < 6 Months vs Placebo and Cytarabine - In Stratum < 6 Months; Participants stratified by calculated strata - CR1 <6 months [Complete Remission (CR)]; Test type: Superiority or Other; p = 0.0353, Fisher Exact
Statistical Analysis 6: Comparison: Clofarabine and Cytarabine In Stratum >= 6 Months vs Placebo and Cytarabine In Stratum >= 6 Months; Participants stratified by calculated strata - CR1 >=6 months [Complete Remission (CR)]; Test type: Superiority or Other; p = 0.0096, Fisher Exact

3. Secondary Outcome: Duration of Remission (DOR) Per IRRP Assessment-Overall and by Calculated Strata (CSR 7-April-11)
Description: DOR was defined as the time from first CR or CRi to the date of first objective documentation of disease recurrence, initiation of alternative antileukemic therapy [including hematopoietic stem cell transplant] while in remission, or death due to any cause, whichever occurred first.
  CR is defined on morphologic criteria at a single response assessment:
  * a bone marrow aspirate or biopsy of <5% blasts, with evidence of normal hematopoiesis;
  * absence of Auer rods in the blasts that are present;
  * absence of extramedullary disease;
  * absence of a unique phenotype determined at the pretreatment specimen, as assessed by immunophenotyping;
  * only rare evidence of circulating blasts. If present, evidence of a regenerating bone marrow;
  * recovery of peripheral counts (platelets ≥100*10^9/L and absolute neutrophil count (ANC) ≥1.0*10^9/L).
  CRi met all criteria for CR except for either residual neutropenia (ANC <1.0*10^9/L) or thrombocytopenia (platelet count <100*10^9/L).
Time Frame: Day 12 to approximately 4 years
Population: Participants in the FAS who achieved OR (CR + CRi). Strata are calculated according to duration of the first remission based on case report forms (CRF) data and do not include the IVRS mistakes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine | Clofarabine and Cytarabine - In Stratum < 6 Months | Placebo and Cytarabine - In Stratum < 6 Months | Clofarabine and Cytarabine In Stratum >= 6 Months | Placebo and Cytarabine In Stratum >= 6 Months
Number analyzed (Participants) | 76 | 36 | 40 | 19 | 36 | 17
months | 7.6 [5.4 to 11.5] | 3.8 [3.3 to 12.1] | 5.7 [5.3 to 7.7] | 6.3 [2.3 to 7.2] | 11.5 [6.8 to 15.5] | 3.8 [3.3 to NA] — N/A = There were an insufficient number of events to allow estimation of the upper limit.

4. Secondary Outcome: Duration of Remission (DOR) Per IRRP Assessment-Overall and by Randomized Strata (CSR 9-July-12)
Description: as for outcome 3
Time Frame: Day 12 to approximately 4 years
Population: Participants in the FAS who achieved OR (CR + CRi). Strata are as randomized by the IVRS, therefore strata include the IVRS mistakes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine | Clofarabine and Cytarabine - In Stratum < 6 Months | Placebo and Cytarabine - In Stratum < 6 Months | Clofarabine and Cytarabine In Stratum >= 6 Months | Placebo and Cytarabine In Stratum >= 6 Months
Number analyzed (Participants) | 76 | 36 | 36 | 20 | 40 | 16
months | 7.7 [5.7 to 11.5] | 3.8 [3.3 to 12.1] | 6.7 [4.0 to 8.8] | 6.3 [2.3 to 7.2] | 10.2 [6.8 to 20.2] | 3.8 [3.3 to NA] — There were an insufficient number of events to allow estimation of the upper limit.

5. Secondary Outcome: Disease-free Survival by IRRP Assessment - Overall and by Calculated Strata (CSR 7-April-11)
Description: Disease-free survival was defined as the time from first complete remission (CR) or complete remission with incomplete peripheral blood count recovery (CRi) until the date of first objective documentation of disease recurrence or death due to any cause, whichever occurred first.
  See Outcome #3 for definition of CR and CRi.
  Disease recurrence - reappearance of leukemic blasts in the peripheral blood, confirmed by ≥5% blasts in the bone marrow, and reappearance or development of pathologically proven extramedullary disease.
Time Frame: Day 12 to approximately 4 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine | Clofarabine and Cytarabine - In Stratum < 6 Months | Placebo and Cytarabine - In Stratum < 6 Months | Clofarabine and Cytarabine In Stratum >= 6 Months | Placebo and Cytarabine In Stratum >= 6 Months
Number analyzed (Participants) | 76 | 36 | 40 | 19 | 36 | 17
months | 8.1 [6.7 to 10.3] | 7.0 [3.9 to 12.1] | 5.7 [4.4 to 9.7] | 6.7 [3.9 to 8.1] | 10.3 [7.5 to 15.5] | 9.1 [3.7 to NA] — NA = There were an insufficient number of events to allow estimation of the upper limit.

6. Secondary Outcome: Disease-free Survival by IRRP Assessment - Overall and by Randomized Strata (CSR 9-July-12)
Description: as for outcome 5
Time Frame: Day 12 to approximately 4 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine | Clofarabine and Cytarabine - In Stratum < 6 Months | Placebo and Cytarabine - In Stratum < 6 Months | Clofarabine and Cytarabine In Stratum >= 6 Months | Placebo and Cytarabine In Stratum >= 6 Months
Number analyzed (Participants) | 76 | 36 | 36 | 20 | 40 | 16
months | 9.5 [6.9 to 15.4] | 7.0 [3.9 to 9.8] | 6.7 [3.9 to 9.7] | 6.7 [3.9 to 8.1] | 15.4 [9.2 to 20.5] | 9.2 [3.7 to 13.1]

7. Secondary Outcome: Event-free Survival by IRRP Assessment - Overall and by Calculated Strata (CSR 7-April-11)
Description: Event-free survival (EFS) was defined as the time from randomization to the date of treatment failure, first disease recurrence (for participants who achieved remission), or death due to any cause, whichever occurred first.
  Treatment Failure - ≥5% leukemic blasts by bone marrow exam, with no evidence of hematologic response (ie, <30% decrease in % leukemic blasts).
  Disease recurrence - reappearance of leukemic blasts in the peripheral blood, confirmed by ≥5% blasts in the bone marrow, and reappearance or development of pathologically proven extramedullary disease.
Time Frame: Day 1 (randomization) up to approximately 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine | Clofarabine and Cytarabine - In Stratum < 6 Months | Placebo and Cytarabine - In Stratum < 6 Months | Clofarabine and Cytarabine In Stratum >= 6 Months | Placebo and Cytarabine In Stratum >= 6 Months
Number analyzed (Participants) | 162 | 157 | 88 | 83 | 74 | 74
months | 1.9 [1.1 to 2.9] | 1.0 [0.9 to 1.1] | 1.4 [1.0 to 2.9] | 1.0 [0.7 to 1.2] | 2.0 [1.2 to 6.6] | 1.0 [0.9 to 1.2]
Statistical Analysis 1: Comparison: Clofarabine (IV Formulation) and Cytarabine vs Placebo and Cytarabine; Full Analysis Set (FAS) population; Test type: Superiority or Other; p = 0.0001, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.49 to 0.80]
Statistical Analysis 2: Comparison: Clofarabine and Cytarabine - In Stratum < 6 Months vs Placebo and Cytarabine - In Stratum < 6 Months; Participants stratified by randomization strata CR1 <6 months; Test type: Superiority or Other; p = 0.0131, Log Rank; Comparison P-value is from a log-rank test with no strata; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.49 to 0.93]
Statistical Analysis 3: Comparison: Clofarabine and Cytarabine In Stratum >= 6 Months vs Placebo and Cytarabine In Stratum >= 6 Months; Participants stratified by randomization strata CR1 >=6 months; Test type: Superiority or Other; p = 0.0022, Log Rank; Comparison p-value is from a log-rank test with no strata; Hazard Ratio (HR) = 0.57, 95% CI [0.40 to 0.83]

8. Primary Outcome: Overall Survival - Overall and by Randomized Strata (CSR 9-July-12)
Description: Overall survival (OS) for the Full Analysis Set (FAS) and for the 2 randomized strata. OS was defined as the number of months from date of randomization until date of death due to any cause.
Time Frame: Day 1 (randomization) up to approximately 4 years
Population: Full Analysis Set (FAS) - composed of all randomized participants whose baseline AML diagnosis was centrally confirmed. Strata are as randomized by the IVRS, therefore strata include the IVRS mistakes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clofarabine (IV Formulation) and Cytarabine (FAS) | Placebo and Cytarabine (FAS) | Clofarabine and Cytarabine - In Stratum < 6 Months | Placebo and Cytarabine - In Stratum < 6 Months | Clofarabine and Cytarabine In Stratum >= 6 Months | Placebo and Cytarabine In Stratum >= 6 Months
Number analyzed (Participants) | 162 | 158 | 86 | 84 | 76 | 74
months | 6.6 [5.1 to 9.3] | 6.3 [4.7 to 7.3] | 4.8 [2.9 to 7.3] | 6.3 [4.1 to 7.8] | 9.7 [5.9 to 12.7] | 6.6 [4.3 to 8.8]
Statistical Analysis 1: Comparison: Clofarabine (IV Formulation) and Cytarabine (FAS) vs Placebo and Cytarabine (FAS); Full Analysis Set (FAS) population; Test type: Superiority or Other; p = 0.8209, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.77 to 1.23]
Statistical Analysis 2: Comparison: Clofarabine and Cytarabine - In Stratum < 6 Months vs Placebo and Cytarabine - In Stratum < 6 Months; Test type: Superiority or Other; p = 0.5071, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.81 to 1.53]
Statistical Analysis 3: Comparison: Clofarabine and Cytarabine In Stratum >= 6 Months vs Placebo and Cytarabine In Stratum >= 6 Months; Test type: Superiority or Other; p = 0.2906, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.59 to 1.17]

9. Secondary Outcome: Event-free Survival by IRRP Assessment - Overall and by Randomized Strata (CSR 9-July-12)
Description: as for outcome 7
Time Frame: Day 1 (randomization) up to approximately 4 years
Population: Full Analysis Set - composed of all randomized participants whose baseline AML diagnosis was centrally confirmed. Strata are as randomized by the IVRS, therefore strata include the IVRS mistakes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine | Clofarabine and Cytarabine - In Stratum < 6 Months | Placebo and Cytarabine - In Stratum < 6 Months | Clofarabine and Cytarabine In Stratum >= 6 Months | Placebo and Cytarabine In Stratum >= 6 Months
Number analyzed (Participants) | 162 | 158 | 86 | 84 | 76 | 74
months | 1.9 [1.1 to 2.9] | 1.0 [0.8 to 1.1] | 1.1 [0.8 to 2.5] | 1.0 [0.7 to 1.2] | 2.8 [1.2 to 8.1] | 1.0 [0.8 to 1.2]
Statistical Analysis 1: Comparison: Clofarabine (IV Formulation) and Cytarabine vs Placebo and Cytarabine; Full Analysis Set (FAS) population; Test type: Superiority or Other; p < .0001, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.49 to 0.79]
Statistical Analysis 2: Comparison: Clofarabine and Cytarabine - In Stratum < 6 Months vs Placebo and Cytarabine - In Stratum < 6 Months; Test type: Superiority or Other; p = 0.0486, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.53 to 1.01]
Statistical Analysis 3: Comparison: Clofarabine and Cytarabine In Stratum >= 6 Months vs Placebo and Cytarabine In Stratum >= 6 Months; Test type: Superiority or Other; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.37 to 0.74]

10. Secondary Outcome: Four-Month Event-free Survival Per IRRP Assessment - Overall and by Calculated Strata (CSR 7-April-11)
Description: Four-month event-free survival (EFS) was defined as achieving an EFS of at least 122 days, where EFS is defined as the time from randomization to the date of treatment failure, first disease recurrence (for participants who achieved remission), or death due to any cause, whichever occurred first.
  Treatment Failure - ≥5% leukemic blasts by bone marrow exam, with no evidence of hematologic response (ie, <30% decrease in % leukemic blasts).
  Disease recurrence - reappearance of leukemic blasts in the peripheral blood, confirmed by ≥5% blasts in the bone marrow, and reappearance or development of pathologically proven extramedullary disease.
Time Frame: Day 1 (randomization) to Day 122
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine | Clofarabine and Cytarabine - In Stratum < 6 Months | Placebo and Cytarabine - In Stratum < 6 Months | Clofarabine and Cytarabine In Stratum >= 6 Months | Placebo and Cytarabine In Stratum >= 6 Months
Number analyzed (Participants) | 162 | 157 | 88 | 83 | 74 | 74
percentage of participants | 37.7 | 16.6 | 35.2 | 16.9 | 40.5 | 16.2
Statistical Analysis 1: Comparison: Clofarabine (IV Formulation) and Cytarabine vs Placebo and Cytarabine; Full Analysis Set (FAS) population; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Clofarabine and Cytarabine - In Stratum < 6 Months vs Placebo and Cytarabine - In Stratum < 6 Months; Participants stratified by randomization strata CR1 <6 months; Test type: Superiority or Other; p = 0.0088, Fisher Exact
Statistical Analysis 3: Comparison: Clofarabine and Cytarabine In Stratum >= 6 Months vs Placebo and Cytarabine In Stratum >= 6 Months; Participants stratified by randomization strata CR1 >=6 months; Test type: Superiority or Other; p = 0.0017, Fisher Exact

11. Secondary Outcome: Four-Month Event-free Survival Per IRRP Assessment - Overall and by Randomized Strata (CSR 9-July-12)
Description: as for outcome 10
Time Frame: Day 1 (randomization) to Day 122
Population: Full Analysis Set - composed of all randomized participants whose baseline AML diagnosis was centrally confirmed. Strata are as randomized by the IVRS, that is the strata include the IVRS mistakes.
Measure: Number; unit: percentage of participants
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine | Clofarabine and Cytarabine - In Stratum < 6 Months | Placebo and Cytarabine - In Stratum < 6 Months | Clofarabine and Cytarabine In Stratum >= 6 Months | Placebo and Cytarabine In Stratum >= 6 Months
Number analyzed (Participants) | 162 | 158 | 86 | 84 | 76 | 74
percentage of participants | 38.9 | 17.1 | 31.4 | 17.9 | 47.4 | 16.2
Statistical Analysis 1: Comparison: Clofarabine (IV Formulation) and Cytarabine vs Placebo and Cytarabine; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Clofarabine and Cytarabine - In Stratum < 6 Months vs Placebo and Cytarabine - In Stratum < 6 Months; Test type: Superiority or Other; p = 0.0506, Fisher Exact
Statistical Analysis 3: Comparison: Clofarabine and Cytarabine In Stratum >= 6 Months vs Placebo and Cytarabine In Stratum >= 6 Months; Test type: Superiority or Other; p < 0.0001, Fisher Exact

12. Secondary Outcome: Participants With Adverse Events (CSR 7-April-11)
Description: Number of participants with treatment emergent adverse events (TEAEs) or death due to related AE. Related AEs for the combination arm can be related to either clofarabine or cytarabine.
  Grade 1 = Mild AE, Grade 2 = Moderate AE, Grade 3 = Severe AE, Grade 4 = Life Threatening AE, Grade 5 = Death
Time Frame: Day 1 up to a maximum of 4 years (includes up to a maximum of 3 cycles of therapy plus 45 days follow up. Related AEs are followed to resolution.)
Population: Safety Set - Participants in the Full Analysis Set (FAS) who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine
Number analyzed (Participants) | 161 | 155
participants
  Any Treatment Emergent AE | 161 | 155
  Any Related Treatment Emergent AE | 157 | 133
  Any Treatment Emergent Grade >=3 AE | 157 | 133
  Any Related Treatment Related Grade >=3 AE | 127 | 83
  Discontinue of study medication due to AE | 17 | 5
  Discontinue of study medication due to related AE | 14 | 3

ADVERSE EVENTS:
Time Frame: Day 1 up to a maximum of 4 years (includes up to a maximum of 3 cycles of therapy plus 45 days follow up. Related AEs are followed to resolution.)
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. Adverse event information is from the final database supporting the clinical study report dated 9-July-12.
Groups:
- Overall: Combined total for the two Arms/Groups
Arm/Group | Clofarabine (IV Formulation) and Cytarabine | Placebo and Cytarabine | Overall
Serious Adverse Events (participants affected / at risk) | 97/161 | 76/155 | 173/316
Other Adverse Events (participants affected / at risk) | 161/161 | 154/155 | 315/316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clofarabine (IV Formulation) and Cytarabine (N=161) | Placebo and Cytarabine (N=155) | Overall (N=316)
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 25 | 19 | 44
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 6
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 5
Acute myocardial infarction (Cardiac disorders) | 3 | 0 | 3
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 3
Atrial flutter (Cardiac disorders) | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 2 | 3
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Blindness unilateral (Eye disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Caecitis (Gastrointestinal disorders) | 0 | 2 | 2
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 3 | 1 | 4
Death (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 1
Hypothermia (General disorders) | 0 | 1 | 1
Inflammation (General disorders) | 0 | 1 | 1
Multi-organ failure (General disorders) | 3 | 1 | 4
Oedema peripheral (General disorders) | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 7 | 9 | 16
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Graft versus host disease (Immune system disorders) | 0 | 1 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 7 | 3 | 10
Bacterial infection (Infections and infestations) | 0 | 1 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 1 | 3
Cellulitis (Infections and infestations) | 0 | 3 | 3
Clostridial infection (Infections and infestations) | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 3 | 2 | 5
Corynebacterium sepsis (Infections and infestations) | 1 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 2 | 2
Enterobacter sepsis (Infections and infestations) | 1 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 6 | 1 | 7
Enterococcal sepsis (Infections and infestations) | 3 | 0 | 3
Escherichia bacteraemia (Infections and infestations) | 4 | 0 | 4
Escherichia infection (Infections and infestations) | 0 | 1 | 1
Escherichia sepsis (Infections and infestations) | 2 | 0 | 2
Fungal infection (Infections and infestations) | 1 | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Keratitis herpetic (Infections and infestations) | 1 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 2 | 2
Lobar pneumonia (Infections and infestations) | 0 | 1 | 1
Neutropenic sepsis (Infections and infestations) | 4 | 0 | 4
Oral herpes (Infections and infestations) | 1 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 13 | 12 | 25
Pneumonia bacterial (Infections and infestations) | 3 | 0 | 3
Pneumonia fungal (Infections and infestations) | 5 | 0 | 5
Pneumonia viral (Infections and infestations) | 0 | 1 | 1
Pseudomonal bacteraemia (Infections and infestations) | 1 | 1 | 2
Sepsis (Infections and infestations) | 8 | 3 | 11
Sepsis syndrome (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 6 | 0 | 6
Serratia sepsis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 2 | 2 | 4
Staphylococcal infection (Infections and infestations) | 1 | 1 | 2
Staphylococcal scalded skin syndrome (Infections and infestations) | 1 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 0 | 2
Streptococcal bacteraemia (Infections and infestations) | 4 | 0 | 4
Streptococcal sepsis (Infections and infestations) | 2 | 0 | 2
Systemic candida (Infections and infestations) | 1 | 0 | 1
Upper respiratory fungal infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 2 | 3
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 1
Zygomycosis (Infections and infestations) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Blood phosphorus decreased (Investigations) | 1 | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 1
Troponin I increased (Investigations) | 1 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 9
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 6
Cerebral haemorrhage (Nervous system disorders) | 2 | 2 | 4
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 2
Convulsion (Nervous system disorders) | 1 | 1 | 2
Encephalopathy (Nervous system disorders) | 1 | 1 | 2
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 2 | 0 | 2
Agitation (Psychiatric disorders) | 1 | 1 | 2
Confusional state (Psychiatric disorders) | 0 | 2 | 2
Mental status changes (Psychiatric disorders) | 1 | 1 | 2
Anuria (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 5 | 1 | 6
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 1
Renal infarct (Renal and urinary disorders) | 0 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 3
Hypertension (Vascular disorders) | 0 | 2 | 2
Hypotension (Vascular disorders) | 4 | 4 | 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clofarabine (IV Formulation) and Cytarabine (N=161) | Placebo and Cytarabine (N=155) | Overall (N=316)
Anaemia (Blood and lymphatic system disorders) | 26 | 18 | 44
Coagulopathy (Blood and lymphatic system disorders) | 10 | 1 | 11
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0 | 2
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 58 | 35 | 93
Haemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1 | 1
Hyperfibrinogenaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 9 | 7 | 16
Lymph node pain (Blood and lymphatic system disorders) | 2 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 5 | 8
Lymphatic disorder (Blood and lymphatic system disorders) | 0 | 1 | 1
Monocytosis (Blood and lymphatic system disorders) | 1 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 17 | 10 | 27
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0 | 3
Splenomegaly (Blood and lymphatic system disorders) | 1 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 23 | 50
Angina pectoris (Cardiac disorders) | 5 | 2 | 7
Aortic valve calcification (Cardiac disorders) | 1 | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 2 | 3 | 5
Arrhythmia supraventricular (Cardiac disorders) | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 6 | 3 | 9
Atrial flutter (Cardiac disorders) | 5 | 0 | 5
Atrioventricular block (Cardiac disorders) | 2 | 0 | 2
Atrioventricular block first degree (Cardiac disorders) | 3 | 0 | 3
Bradycardia (Cardiac disorders) | 3 | 14 | 17
Bundle branch block left (Cardiac disorders) | 2 | 1 | 3
Bundle branch block right (Cardiac disorders) | 3 | 0 | 3
Cardiac aneurysm (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 2
Cardiac valve disease (Cardiac disorders) | 1 | 1 | 2
Cardiomegaly (Cardiac disorders) | 4 | 0 | 4
Conduction disorder (Cardiac disorders) | 1 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 2 | 0 | 2
Dilatation atrial (Cardiac disorders) | 0 | 1 | 1
Dilatation ventricular (Cardiac disorders) | 0 | 1 | 1
Extrasystoles (Cardiac disorders) | 1 | 0 | 1
Heart valve incompetence (Cardiac disorders) | 1 | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Left atrial dilatation (Cardiac disorders) | 2 | 1 | 3
Left ventricular dysfunction (Cardiac disorders) | 1 | 2 | 3
Left ventricular hypertrophy (Cardiac disorders) | 2 | 1 | 3
Mitral valve incompetence (Cardiac disorders) | 4 | 3 | 7
Myocardial infarction (Cardiac disorders) | 1 | 4 | 5
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 2 | 3 | 5
Pericardial effusion (Cardiac disorders) | 3 | 6 | 9
Pulmonary valve incompetence (Cardiac disorders) | 1 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 3 | 0 | 3
Sinus bradycardia (Cardiac disorders) | 3 | 2 | 5
Sinus tachycardia (Cardiac disorders) | 12 | 6 | 18
Supraventricular extrasystoles (Cardiac disorders) | 1 | 3 | 4
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 25 | 14 | 39
Tricuspid valve incompetence (Cardiac disorders) | 3 | 3 | 6
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 4 | 2 | 6
Ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 1
Ventricular hypokinesia (Cardiac disorders) | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 3 | 5
Hypoacusis (Ear and labyrinth disorders) | 2 | 1 | 3
Tinnitus (Ear and labyrinth disorders) | 2 | 2 | 4
Vertigo (Ear and labyrinth disorders) | 4 | 2 | 6
Adrenal disorder (Endocrine disorders) | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 1
Cushingoid (Endocrine disorders) | 1 | 0 | 1
Hyperadrenalism (Endocrine disorders) | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
Thyroid mass (Endocrine disorders) | 0 | 1 | 1
Blepharitis (Eye disorders) | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Conjunctival cyst (Eye disorders) | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 5 | 3 | 8
Conjunctival hyperaemia (Eye disorders) | 2 | 1 | 3
Conjunctival pallor (Eye disorders) | 2 | 0 | 2
Conjunctivitis (Eye disorders) | 1 | 1 | 2
Diplopia (Eye disorders) | 1 | 0 | 1
Dry eye (Eye disorders) | 7 | 7 | 14
Erythema of eyelid (Eye disorders) | 1 | 1 | 2
Eye haemorrhage (Eye disorders) | 2 | 1 | 3
Eye irritation (Eye disorders) | 3 | 2 | 5
Eye pain (Eye disorders) | 3 | 2 | 5
Eye swelling (Eye disorders) | 1 | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 2 | 3
Eyelid ptosis (Eye disorders) | 1 | 0 | 1
Gaze palsy (Eye disorders) | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 2 | 0 | 2
Miosis (Eye disorders) | 1 | 0 | 1
Ocular dysmetria (Eye disorders) | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 2 | 2
Ocular icterus (Eye disorders) | 1 | 0 | 1
Optic neuropathy (Eye disorders) | 2 | 0 | 2
Papilloedema (Eye disorders) | 1 | 0 | 1
Periorbital oedema (Eye disorders) | 4 | 1 | 5
Photophobia (Eye disorders) | 3 | 1 | 4
Pupillary reflex impaired (Eye disorders) | 0 | 2 | 2
Pupils unequal (Eye disorders) | 2 | 0 | 2
Retinal haemorrhage (Eye disorders) | 1 | 0 | 1
Scleral disorder (Eye disorders) | 1 | 0 | 1
Scleral haemorrhage (Eye disorders) | 1 | 0 | 1
Scleral oedema (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 8 | 4 | 12
Visual acuity reduced (Eye disorders) | 1 | 0 | 1
Visual impairment (Eye disorders) | 1 | 1 | 2
Vitreous detachment (Eye disorders) | 0 | 1 | 1
Vitreous floaters (Eye disorders) | 1 | 2 | 3
Abdominal discomfort (Gastrointestinal disorders) | 5 | 3 | 8
Abdominal distension (Gastrointestinal disorders) | 18 | 13 | 31
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 30 | 18 | 48
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 6 | 11
Abdominal tenderness (Gastrointestinal disorders) | 3 | 2 | 5
Anal inflammation (Gastrointestinal disorders) | 1 | 1 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 3 | 1 | 4
Caecitis (Gastrointestinal disorders) | 2 | 0 | 2
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 1 | 3
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 1
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 66 | 72 | 138
Crohn's disease (Gastrointestinal disorders) | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 109 | 63 | 172
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 9 | 6 | 15
Dyspepsia (Gastrointestinal disorders) | 12 | 19 | 31
Dysphagia (Gastrointestinal disorders) | 7 | 4 | 11
Epigastric discomfort (Gastrointestinal disorders) | 2 | 0 | 2
Eructation (Gastrointestinal disorders) | 0 | 1 | 1
Faecal incontinence (Gastrointestinal disorders) | 5 | 5 | 10
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 10 | 4 | 14
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 3
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 5 | 7
Gingival bleeding (Gastrointestinal disorders) | 5 | 2 | 7
Gingival cyst (Gastrointestinal disorders) | 0 | 1 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 1 | 2
Gingivitis (Gastrointestinal disorders) | 6 | 1 | 7
Glossodynia (Gastrointestinal disorders) | 0 | 3 | 3
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 2
Haematochezia (Gastrointestinal disorders) | 5 | 3 | 8
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 3
Haemorrhoids (Gastrointestinal disorders) | 13 | 9 | 22
Hiatus hernia (Gastrointestinal disorders) | 2 | 1 | 3
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 1 | 3
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal dilatation (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Lip blister (Gastrointestinal disorders) | 1 | 1 | 2
Lip dry (Gastrointestinal disorders) | 4 | 5 | 9
Lip haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 1 | 1 | 2
Melaena (Gastrointestinal disorders) | 1 | 2 | 3
Mouth haemorrhage (Gastrointestinal disorders) | 11 | 7 | 18
Mouth ulceration (Gastrointestinal disorders) | 3 | 9 | 12
Mucous stools (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 117 | 82 | 199
Neutropenic colitis (Gastrointestinal disorders) | 2 | 0 | 2
Odynophagia (Gastrointestinal disorders) | 1 | 1 | 2
Oesophageal dilatation (Gastrointestinal disorders) | 0 | 1 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 2 | 1 | 3
Oral disorder (Gastrointestinal disorders) | 2 | 4 | 6
Oral mucosal discolouration (Gastrointestinal disorders) | 1 | 3 | 4
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 2 | 3
Oral pain (Gastrointestinal disorders) | 2 | 1 | 3
Pancreatic mass (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 2
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0 | 1
Poor dental condition (Gastrointestinal disorders) | 1 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 2 | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 4 | 6
Rectal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Retching (Gastrointestinal disorders) | 3 | 1 | 4
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 17 | 10 | 27
Tongue blistering (Gastrointestinal disorders) | 0 | 1 | 1
Tongue coated (Gastrointestinal disorders) | 0 | 1 | 1
Tongue discolouration (Gastrointestinal disorders) | 2 | 4 | 6
Tongue exfoliation (Gastrointestinal disorders) | 0 | 1 | 1
Tongue haematoma (Gastrointestinal disorders) | 1 | 2 | 3
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 8 | 3 | 11
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 71 | 42 | 113
Adverse event (General disorders) | 1 | 0 | 1
Asthenia (General disorders) | 32 | 33 | 65
Catheter site discharge (General disorders) | 1 | 0 | 1
Catheter site erosion (General disorders) | 1 | 0 | 1
Catheter site erythema (General disorders) | 6 | 13 | 19
Catheter site haematoma (General disorders) | 4 | 0 | 4
Catheter site haemorrhage (General disorders) | 6 | 4 | 10
Catheter site inflammation (General disorders) | 2 | 0 | 2
Catheter site oedema (General disorders) | 1 | 1 | 2
Catheter site pain (General disorders) | 12 | 9 | 21
Catheter site pruritus (General disorders) | 1 | 0 | 1
Catheter site rash (General disorders) | 1 | 2 | 3
Catheter site related reaction (General disorders) | 2 | 5 | 7
Catheter site swelling (General disorders) | 1 | 2 | 3
Chest discomfort (General disorders) | 4 | 4 | 8
Chest pain (General disorders) | 3 | 2 | 5
Chills (General disorders) | 38 | 23 | 61
Crepitations (General disorders) | 1 | 0 | 1
Cyst (General disorders) | 0 | 1 | 1
Device occlusion (General disorders) | 3 | 1 | 4
Discomfort (General disorders) | 0 | 1 | 1
Early satiety (General disorders) | 1 | 0 | 1
Face oedema (General disorders) | 2 | 2 | 4
Facial pain (General disorders) | 1 | 2 | 3
Fatigue (General disorders) | 57 | 49 | 106
Feeling cold (General disorders) | 1 | 1 | 2
Feeling hot (General disorders) | 0 | 1 | 1
Gait disturbance (General disorders) | 2 | 1 | 3
General physical health deterioration (General disorders) | 3 | 2 | 5
Generalised oedema (General disorders) | 9 | 4 | 13
Hypothermia (General disorders) | 1 | 0 | 1
Infusion site discolouration (General disorders) | 1 | 0 | 1
Infusion site induration (General disorders) | 1 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 1 | 1
Injection site inflammation (General disorders) | 0 | 1 | 1
Injection site pain (General disorders) | 1 | 0 | 1
Injection site reaction (General disorders) | 4 | 1 | 5
Malaise (General disorders) | 2 | 2 | 4
Mass (General disorders) | 1 | 0 | 1
Medical device complication (General disorders) | 0 | 1 | 1
Mucosal dryness (General disorders) | 0 | 1 | 1
Mucosal inflammation (General disorders) | 21 | 19 | 40
Nodule (General disorders) | 1 | 1 | 2
Non-cardiac chest pain (General disorders) | 6 | 3 | 9
Oedema (General disorders) | 4 | 5 | 9
Oedema peripheral (General disorders) | 82 | 71 | 153
Pain (General disorders) | 22 | 8 | 30
Pyrexia (General disorders) | 53 | 39 | 92
Tenderness (General disorders) | 1 | 2 | 3
Thrombosis in device (General disorders) | 3 | 1 | 4
Visceral oedema (General disorders) | 1 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 4 | 8
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 1 | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 2 | 2 | 4
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 2 | 0 | 2
Hepatic steatosis (Hepatobiliary disorders) | 2 | 2 | 4
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 3 | 3
Hepatosplenomegaly (Hepatobiliary disorders) | 2 | 0 | 2
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 15 | 12 | 27
Jaundice (Hepatobiliary disorders) | 2 | 0 | 2
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 9 | 1 | 10
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 | 1 | 2
Anal abscess (Infections and infestations) | 1 | 1 | 2
Anorectal infection (Infections and infestations) | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 8 | 4 | 12
Bacterial infection (Infections and infestations) | 1 | 1 | 2
Bacterial sepsis (Infections and infestations) | 1 | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 2 | 3
Bullous impetigo (Infections and infestations) | 1 | 0 | 1
Candida pneumonia (Infections and infestations) | 0 | 1 | 1
Candidiasis (Infections and infestations) | 6 | 3 | 9
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 1
Catheter site infection (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 5 | 9 | 14
Clostridial infection (Infections and infestations) | 3 | 1 | 4
Clostridium difficile colitis (Infections and infestations) | 5 | 3 | 8
Cystitis (Infections and infestations) | 2 | 0 | 2
Cystitis bacterial (Infections and infestations) | 0 | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0 | 1
Device related infection (Infections and infestations) | 6 | 5 | 11
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 2 | 4
Enterobacter bacteraemia (Infections and infestations) | 2 | 0 | 2
Enterococcal bacteraemia (Infections and infestations) | 9 | 3 | 12
Enterococcal infection (Infections and infestations) | 4 | 2 | 6
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 2 | 2 | 4
Escherichia infection (Infections and infestations) | 1 | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 1 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 1
Eye infection (Infections and infestations) | 0 | 1 | 1
Eye infection fungal (Infections and infestations) | 0 | 1 | 1
Eye infection staphylococcal (Infections and infestations) | 0 | 1 | 1
Folliculitis (Infections and infestations) | 1 | 6 | 7
Fungal infection (Infections and infestations) | 0 | 1 | 1
Fungal skin infection (Infections and infestations) | 0 | 1 | 1
Furuncle (Infections and infestations) | 3 | 1 | 4
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Genital herpes (Infections and infestations) | 1 | 0 | 1
Hepatosplenic candidiasis (Infections and infestations) | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 2 | 4 | 6
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 4 | 1 | 5
Lobar pneumonia (Infections and infestations) | 1 | 1 | 2
Localised infection (Infections and infestations) | 1 | 2 | 3
Lung infection (Infections and infestations) | 3 | 1 | 4
Lung infection pseudomonal (Infections and infestations) | 1 | 0 | 1
Micrococcus infection (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 10 | 8 | 18
Oral fungal infection (Infections and infestations) | 1 | 0 | 1
Oral herpes (Infections and infestations) | 9 | 4 | 13
Osteomyelitis (Infections and infestations) | 2 | 0 | 2
Otitis externa (Infections and infestations) | 1 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 14 | 9 | 23
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1
Pneumonia fungal (Infections and infestations) | 5 | 2 | 7
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 2 | 0 | 2
Pseudomonas infection (Infections and infestations) | 0 | 1 | 1
Pulmonary mycosis (Infections and infestations) | 2 | 3 | 5
Respiratory syncytial virus infection (Infections and infestations) | 2 | 1 | 3
Rhinitis (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 2 | 1 | 3
Septic embolus (Infections and infestations) | 2 | 0 | 2
Serratia bacteraemia (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 2 | 4
Sinusitis fungal (Infections and infestations) | 1 | 0 | 1
Skin candida (Infections and infestations) | 1 | 0 | 1
Skin infection (Infections and infestations) | 1 | 1 | 2
Staphylococcal bacteraemia (Infections and infestations) | 9 | 15 | 24
Staphylococcal infection (Infections and infestations) | 4 | 1 | 5
Staphylococcal scalded skin syndrome (Infections and infestations) | 1 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 3 | 1 | 4
Staphylococcal skin infection (Infections and infestations) | 0 | 1 | 1
Stenotrophomonas infection (Infections and infestations) | 0 | 1 | 1
Streptococcal bacteraemia (Infections and infestations) | 3 | 4 | 7
Streptococcal sepsis (Infections and infestations) | 2 | 0 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 1 | 2
Tooth abscess (Infections and infestations) | 0 | 3 | 3
Tooth infection (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 6
Urinary tract infection (Infections and infestations) | 3 | 0 | 3
Urinary tract infection bacterial (Infections and infestations) | 2 | 3 | 5
Urinary tract infection enterococcal (Infections and infestations) | 4 | 1 | 5
Urinary tract infection pseudomonal (Infections and infestations) | 2 | 0 | 2
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 1 | 1
Viral skin infection (Infections and infestations) | 0 | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 1
Anal injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 12 | 17 | 29
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Eschar (Injury, poisoning and procedural complications) | 0 | 2 | 2
Excoriation (Injury, poisoning and procedural complications) | 9 | 3 | 12
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 1 | 6
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 5 | 5 | 10
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Nail injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 2
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 3 | 3
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 2 | 4
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 1 | 4
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 12 | 19 | 31
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3
Transfusion reaction (Injury, poisoning and procedural complications) | 9 | 7 | 16
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Urethral injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 40 | 13 | 53
Ammonia increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 36 | 8 | 44
Bacterial test (Investigations) | 0 | 1 | 1
Bacterial test positive (Investigations) | 2 | 2 | 4
Blast cells present (Investigations) | 0 | 1 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 11 | 6 | 17
Blood amylase increased (Investigations) | 9 | 2 | 11
Blood beta-D-glucan increased (Investigations) | 0 | 1 | 1
Blood bicarbonate decreased (Investigations) | 5 | 0 | 5
Blood bicarbonate increased (Investigations) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 12 | 1 | 13
Blood calcium decreased (Investigations) | 0 | 1 | 1
Blood chloride decreased (Investigations) | 2 | 0 | 2
Blood chloride increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 6 | 3 | 9
Blood culture positive (Investigations) | 1 | 1 | 2
Blood glucose increased (Investigations) | 2 | 2 | 4
Blood iron increased (Investigations) | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 9 | 4 | 13
Blood magnesium decreased (Investigations) | 3 | 0 | 3
Blood magnesium increased (Investigations) | 1 | 0 | 1
Blood osmolarity increased (Investigations) | 1 | 0 | 1
Blood phosphorus decreased (Investigations) | 1 | 1 | 2
Blood phosphorus increased (Investigations) | 1 | 0 | 1
Blood potassium decreased (Investigations) | 2 | 2 | 4
Blood potassium increased (Investigations) | 1 | 0 | 1
Blood pressure increased (Investigations) | 1 | 1 | 2
Blood urea increased (Investigations) | 2 | 3 | 5
Blood uric acid increased (Investigations) | 1 | 0 | 1
Blood urine present (Investigations) | 1 | 1 | 2
Breath sounds abnormal (Investigations) | 5 | 7 | 12
Cardiac murmur (Investigations) | 6 | 9 | 15
Catheter culture positive (Investigations) | 1 | 0 | 1
Clostridium test positive (Investigations) | 0 | 1 | 1
Crystal urine present (Investigations) | 1 | 0 | 1
Culture stool positive (Investigations) | 1 | 2 | 3
Culture throat positive (Investigations) | 1 | 0 | 1
Culture urine positive (Investigations) | 1 | 0 | 1
Cytomegalovirus test positive (Investigations) | 1 | 0 | 1
Diagnostic procedure (Investigations) | 0 | 1 | 1
Electrocardiogram PR shortened (Investigations) | 1 | 2 | 3
Electrocardiogram QT prolonged (Investigations) | 4 | 5 | 9
Electrocardiogram ST-T segment abnormal (Investigations) | 0 | 2 | 2
Electrocardiogram T wave abnormal (Investigations) | 2 | 1 | 3
Electrocardiogram abnormal (Investigations) | 1 | 2 | 3
Enterococcus test positive (Investigations) | 5 | 3 | 8
Escherichia test positive (Investigations) | 0 | 1 | 1
Fungal test positive (Investigations) | 1 | 0 | 1
Gallop rhythm present (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 3
Glucose urine present (Investigations) | 0 | 1 | 1
Haematocrit decreased (Investigations) | 2 | 0 | 2
Haemoglobin decreased (Investigations) | 3 | 1 | 4
Heart rate decreased (Investigations) | 0 | 1 | 1
Heart rate increased (Investigations) | 2 | 0 | 2
Hepatic enzyme increased (Investigations) | 3 | 0 | 3
International normalised ratio increased (Investigations) | 2 | 0 | 2
Lipase increased (Investigations) | 10 | 3 | 13
Liver function test abnormal (Investigations) | 3 | 7 | 10
Liver scan abnormal (Investigations) | 0 | 1 | 1
Lymph node palpable (Investigations) | 0 | 1 | 1
Monocyte count increased (Investigations) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Nitrite urine present (Investigations) | 0 | 1 | 1
Platelet count decreased (Investigations) | 2 | 0 | 2
Protein total decreased (Investigations) | 2 | 0 | 2
Protein total increased (Investigations) | 1 | 0 | 1
Protein urine present (Investigations) | 0 | 1 | 1
Prothrombin time prolonged (Investigations) | 2 | 1 | 3
Pulmonary function test decreased (Investigations) | 1 | 0 | 1
QRS axis abnormal (Investigations) | 1 | 0 | 1
Red blood cell count decreased (Investigations) | 2 | 0 | 2
Red blood cells urine positive (Investigations) | 0 | 1 | 1
Right ventricular systolic pressure increased (Investigations) | 0 | 1 | 1
Serum ferritin increased (Investigations) | 1 | 0 | 1
Spleen palpable (Investigations) | 1 | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 1 | 1
Streptococcus test positive (Investigations) | 2 | 1 | 3
Total lung capacity decreased (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 10 | 1 | 11
Troponin I increased (Investigations) | 1 | 0 | 1
Urinary sediment present (Investigations) | 0 | 1 | 1
Urine leukocyte esterase positive (Investigations) | 1 | 0 | 1
Urine output decreased (Investigations) | 0 | 2 | 2
Weight decreased (Investigations) | 24 | 11 | 35
Weight increased (Investigations) | 13 | 7 | 20
White blood cell count decreased (Investigations) | 2 | 1 | 3
White blood cell count increased (Investigations) | 1 | 0 | 1
White blood cells urine positive (Investigations) | 1 | 0 | 1
pH urine increased (Investigations) | 0 | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 2 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 57 | 37 | 94
Dehydration (Metabolism and nutrition disorders) | 8 | 4 | 12
Diabetes mellitus (Metabolism and nutrition disorders) | 8 | 4 | 12
Fluid overload (Metabolism and nutrition disorders) | 22 | 17 | 39
Fluid retention (Metabolism and nutrition disorders) | 9 | 7 | 16
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 17 | 17 | 34
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 1 | 6
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 | 2 | 4
Hypernatraemia (Metabolism and nutrition disorders) | 4 | 1 | 5
Hyperphosphataemia (Metabolism and nutrition disorders) | 7 | 7 | 14
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 3 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 22 | 8 | 30
Hypocalcaemia (Metabolism and nutrition disorders) | 14 | 5 | 19
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 3 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 61 | 29 | 90
Hypomagnesaemia (Metabolism and nutrition disorders) | 26 | 13 | 39
Hyponatraemia (Metabolism and nutrition disorders) | 15 | 5 | 20
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 12 | 7 | 19
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Iron overload (Metabolism and nutrition disorders) | 1 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 4 | 1 | 5
Metabolic acidosis (Metabolism and nutrition disorders) | 4 | 1 | 5
Polydipsia (Metabolism and nutrition disorders) | 1 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 7 | 23
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 16 | 45
Bone loss (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Chondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 5 | 13
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 | 1 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 9
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 9 | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 7 | 16
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 7 | 12
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 12 | 39
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Benign neoplasm of eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0 | 1
Apraxia (Nervous system disorders) | 1 | 0 | 1
Ataxia (Nervous system disorders) | 2 | 1 | 3
Burning sensation (Nervous system disorders) | 2 | 1 | 3
Carotid arteriosclerosis (Nervous system disorders) | 2 | 0 | 2
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 1
Cerebral atrophy (Nervous system disorders) | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 1
Convulsion (Nervous system disorders) | 3 | 0 | 3
Cranial nerve disorder (Nervous system disorders) | 1 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 19 | 28 | 47
Dizziness postural (Nervous system disorders) | 0 | 1 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 10 | 4 | 14
Dyskinesia (Nervous system disorders) | 1 | 0 | 1
Encephalitis toxic (Nervous system disorders) | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 2 | 3
Headache (Nervous system disorders) | 68 | 44 | 112
Hemiparesis (Nervous system disorders) | 1 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 4 | 7
Hypogeusia (Nervous system disorders) | 1 | 0 | 1
Hypokinesia (Nervous system disorders) | 0 | 1 | 1
Hyporeflexia (Nervous system disorders) | 0 | 1 | 1
Intention tremor (Nervous system disorders) | 1 | 0 | 1
Lethargy (Nervous system disorders) | 3 | 4 | 7
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 1 | 2
Migraine (Nervous system disorders) | 1 | 1 | 2
Myoclonus (Nervous system disorders) | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 4 | 2 | 6
Nystagmus (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 3 | 2 | 5
Peroneal nerve palsy (Nervous system disorders) | 0 | 1 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 2 | 0 | 2
Restless legs syndrome (Nervous system disorders) | 1 | 2 | 3
Sciatica (Nervous system disorders) | 0 | 1 | 1
Sensory disturbance (Nervous system disorders) | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 3 | 4 | 7
Slow speech (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 9 | 7 | 16
Speech disorder (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 6 | 4 | 10
Tension headache (Nervous system disorders) | 1 | 1 | 2
Tremor (Nervous system disorders) | 9 | 7 | 16
Aggression (Psychiatric disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 9 | 2 | 11
Anger (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 35 | 20 | 55
Confusional state (Psychiatric disorders) | 30 | 13 | 43
Delirium (Psychiatric disorders) | 1 | 1 | 2
Depressed mood (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 20 | 8 | 28
Disorientation (Psychiatric disorders) | 0 | 2 | 2
Dysphoria (Psychiatric disorders) | 1 | 0 | 1
Fear (Psychiatric disorders) | 0 | 1 | 1
Flat affect (Psychiatric disorders) | 1 | 1 | 2
Hallucination (Psychiatric disorders) | 3 | 3 | 6
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 51 | 42 | 93
Mental status changes (Psychiatric disorders) | 8 | 4 | 12
Mood altered (Psychiatric disorders) | 1 | 0 | 1
Nightmare (Psychiatric disorders) | 2 | 0 | 2
Panic attack (Psychiatric disorders) | 2 | 0 | 2
Restlessness (Psychiatric disorders) | 2 | 3 | 5
Bladder dilatation (Renal and urinary disorders) | 0 | 1 | 1
Bladder mass (Renal and urinary disorders) | 0 | 1 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 1 | 2
Chromaturia (Renal and urinary disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 8 | 3 | 11
Enuresis (Renal and urinary disorders) | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 8 | 11 | 19
Incontinence (Renal and urinary disorders) | 1 | 0 | 1
Kidney enlargement (Renal and urinary disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Nocturia (Renal and urinary disorders) | 2 | 3 | 5
Oliguria (Renal and urinary disorders) | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 5 | 6 | 11
Polyuria (Renal and urinary disorders) | 1 | 1 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Renal cyst (Renal and urinary disorders) | 4 | 4 | 8
Renal disorder (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 4 | 8
Renal failure acute (Renal and urinary disorders) | 5 | 2 | 7
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 2 | 0 | 2
Urethritis noninfective (Renal and urinary disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 9 | 6 | 15
Urinary retention (Renal and urinary disorders) | 1 | 9 | 10
Urine abnormality (Renal and urinary disorders) | 1 | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 0 | 1 | 1
Balanitis (Reproductive system and breast disorders) | 0 | 1 | 1
Breast haematoma (Reproductive system and breast disorders) | 0 | 1 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 2
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 2 | 0 | 2
Penile blister (Reproductive system and breast disorders) | 1 | 0 | 1
Penile haemorrhage (Reproductive system and breast disorders) | 2 | 2 | 4
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 1
Scrotal oedema (Reproductive system and breast disorders) | 2 | 1 | 3
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 2
Vulvovaginal rash (Reproductive system and breast disorders) | 1 | 0 | 1
Vulvovaginal swelling (Reproductive system and breast disorders) | 1 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 12
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 26 | 60
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 18 | 48
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 30 | 19 | 49
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 16
Hiccups (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 12
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 12
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 10
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 21
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 | 15 | 31
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 10
Rales (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 18
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 6
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 6
Throat lesion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 9
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 3 | 17
Blister (Skin and subcutaneous tissue disorders) | 7 | 3 | 10
Blood blister (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 8 | 1 | 9
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 24 | 13 | 37
Ecchymosis (Skin and subcutaneous tissue disorders) | 9 | 20 | 29
Erythema (Skin and subcutaneous tissue disorders) | 19 | 22 | 41
Exfoliative rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 8
Generalised erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 12 | 6 | 18
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Lentigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 10 | 15
Pain of skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Palmar erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 30 | 2 | 32
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 22 | 24 | 46
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 5 | 24
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Purpura (Skin and subcutaneous tissue disorders) | 2 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 40 | 22 | 62
Rash erythematous (Skin and subcutaneous tissue disorders) | 14 | 3 | 17
Rash follicular (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 17 | 7 | 24
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 4 | 8
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 6 | 1 | 7
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 23 | 3 | 26
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 5 | 8 | 13
Skin mass (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 4 | 5
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 5 | 7
Andropause (Social circumstances) | 1 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 1 | 1 | 2
Aortic calcification (Vascular disorders) | 0 | 2 | 2
Aortic disorder (Vascular disorders) | 1 | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 6 | 3 | 9
Flushing (Vascular disorders) | 19 | 11 | 30
Haematoma (Vascular disorders) | 4 | 3 | 7
Hot flush (Vascular disorders) | 3 | 2 | 5
Hypertension (Vascular disorders) | 29 | 21 | 50
Hypotension (Vascular disorders) | 37 | 33 | 70
Infarction (Vascular disorders) | 1 | 0 | 1
Jugular vein distension (Vascular disorders) | 1 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 2 | 1 | 3
Lymphoedema (Vascular disorders) | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 9 | 4 | 13
Pallor (Vascular disorders) | 2 | 9 | 11
Subclavian vein thrombosis (Vascular disorders) | 1 | 1 | 2
Thrombosis (Vascular disorders) | 3 | 1 | 4
Vascular stenosis (Vascular disorders) | 0 | 1 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 1 | 2
Venous insufficiency (Vascular disorders) | 1 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.